CLINICAL TRIAL: NCT04604002
Title: Evaluation of Additional Heidelberg Engineering SPECTRALIS With OCT Angiography Module (OCTA Module) Scan Types
Acronym: OCTA
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: S-2020-5
Record Dates: First submitted 2020-10-20; First posted 2020-10-27 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Retinal Vascular; Normal Eyes
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Subjects with Normal Eyes: OCT, Color Fundus Photography and OCT Angiography as per protocol in subjects without ophthalmic pathology
  Interventions: Device: OCT Angiography; Device: Color Fundus Photography; Device: Optical Coherence Tomography
- Subjects with Pathology: OCT, Color Fundus Photography and OCT Angiography as per protocol in subjects with retinal vascular pathology
  Interventions: Device: OCT Angiography; Device: Color Fundus Photography; Device: Optical Coherence Tomography

INTERVENTIONS:
Device: OCT Angiography — OCT Angiography offers clinicians a non-invasive three-dimensional visualization of vasculature in the retina and choroid. The visualization of perfused vasculature in a three-dimensional layout, offers clinicians an aid in the identification of retinal and choroidal pathologies such as retinal ischemia, microaneurysms, retinal neovascularization and choroidal neovascular membranes.
  Other Names: Optical Coherence Tomography Angiography; OCTA
Device: Color Fundus Photography — Non-contact white light photography
  Other Names: CFP
Device: Optical Coherence Tomography — A non-contact test that uses light waves to take cross-sectional pictures of the retina
  Other Names: OCT

SUMMARY:
Assessment of image quality and clinical relevance of OCT Angiography at different speed/ART combinations

DETAILED DESCRIPTION:
The objectives of this study are:

1.) Compare the image quality between the predicate scan types and the corresponding investigational scan types.

2. Compare the visibility of key anatomical vascular structures between the predicate scan types and the corresponding investigational scan types.

3. Assess the agreement in identification of vascular abnormalities between the predicate scan types and the corresponding investigational scan types, where agreement is assessed by the vascular abnormalities identified from the predicate scan types.

ELIGIBILITY:
Inclusion Criteria:

* All Populations:

  1. Able and willing to undergo the test procedures, sign informed consent, and follow instructions.
  2. Age ≥ 22
* Normal Population:

  3. Subjects without uncontrolled systemic conditions, as determined by the Investigator 4. Subjects without ocular disease, as determined by the Investigator 5. Corrected visual acuity ≥ 20/40 6. No reported history of ocular surgical intervention (except for refractive or cataract surgery)
* Pathology Population:

  3. Subjects with vascular abnormalities such as retinal ischemia, microaneurysms, choroidal neovascularization, retinal neovascularization in at least one eye

Exclusion Criteria:

* All Populations:

  1. Subjects unable to read or write
  2. Subjects with ocular media not sufficiently clear to obtain acceptable study-related imaging
  3. Subjects who cannot tolerate the imaging procedures
  4. Subjects without an accompanying structural OCT and CFP image for an acceptable OCTA image

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with Healthy Eyes and Adults with Eyes with retinal vascular pathology
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Image quality score | through study completion, an average of 1 day
  Graded 0-2 (0 = poor, 1 = average, 2 = good)
Visibility of OCTA key anatomical vascular structures quality score | through study completion, an average of 1 day
  Graded 0-2 (easy (2), difficult (1) or unable to be distinguished (0)) based on pre-specified abnormalities
Identification of vascular abnormalities on OCTA | through study completion, an average of 1 day
  Graded Yes, No, or Unable to Grade based on pre-specified abnormalities
Adverse Events | through study completion, an average of 1 day
  All AEs

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Marcus, MD, Principal Investigator — Southeast Retina Center
Locations (1):
- Southeast Retina Center, Augusta, Georgia, United States